CLINICAL TRIAL: NCT05890638
Title: A Randomized, Parallel Group, Phase III, Non-inferiority Study Comparing Ipratropium / Levosalbutamol Fixed Dose Combination and Ipratropium and Levosalbutamol Free Dose Combination Nebuliser Solutions in Stable Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Comparison of Ipratropium / Levosalbutamol Fixed Dose Combination and Ipratropium and Levosalbutamol Free Dose Combination Nebuliser Solutions in Stable Chronic Obstructive Pulmonary Disease (COPD) Patients
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Neutec Ar-Ge San ve Tic A.Ş (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NEU-02.22
Record Dates: First submitted 2022-12-23; First posted 2023-06-06 (Actual); Last update posted 2023-09-05 (Actual); Status verified 2023-09

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Ipratropium; Albuterol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ipratropium / Levosalbutamol Fixed Dose Combination (Experimental): In this one-day study, patients will be administered "Ipratropium / Levosalbutamol 1.25 mg & 0.5 mg / 2.5 mL Nebuliser Solution" at 6 hours intervals.
  Interventions: Drug: Ipratropium / Levosalbutamol Fixed Dose Combination
- Ipratropium + Levosalbutamol Free Dose Combination (Active Comparator): In this one-day study, patients will be administered "Levosalbutamol 1.25 mg/3 mL Inhalation Solution" and "Ipratropium Nebulization Solution 500 mcg/2 mL" at 6 hours intervals.
  Interventions: Drug: Ipratropium + Levosalbutamol Free Dose Combination

INTERVENTIONS:
Drug: Ipratropium / Levosalbutamol Fixed Dose Combination — New combination test treatment
  Arms: Ipratropium / Levosalbutamol Fixed Dose Combination
Drug: Ipratropium + Levosalbutamol Free Dose Combination — Free combination control treatment
  Arms: Ipratropium + Levosalbutamol Free Dose Combination

SUMMARY:
The goal of this clinical trial is to compare the acute bronchodilator effect of the Ipratropium / Levosalbutamol 1.25 mg & 0.5 mg / 2.5 mL fixed dose combination nebuliser solution or Levosalbutamol 1.25 mg / 3 mL nebuliser solution and Ipratropium 500 mcg nebuliser solution in stable moderate-severe-very severe COPD patients.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged 40 years and older who have been newly diagnosed or followed up with a diagnosis of COPD.
* Stable moderate-severe-very severe COPD patients with a post-bronchodilator FEV1/FVC ratio <70% and a postbronchodilator FEV1 value <80% at the screening visit will be included in the study.
* Symptom status such as chronic cough, sputum production, and progressive dyspnea with the BCSS (Breathlessness, Cough and Sputum Scale) Index will be evaluated, and the COPD staging of the patient with CAT (COPD Assessment Test) and the severity of dyspnea with mMRC (Modified Medical Research Council) will be determined.
* Patients with at least 10 pack/year smoking status or smoking history (patients who have quit smoking for at least 6 months or more are defined as ex-smokers).
* Patients who have not experienced an exacerbation in the previous 4 weeks.
* If the study participant is female; women using appropriate contraception (pregnancy test will be performed at screening visit).
* Patients with the ability to communicate with the investigator.
* Patients who accept to comply with the protocol.
* Patients who sign written informed consent form.

Exclusion Criteria:

* History of hypersensitivity to anticholinergics or SABAs (short acting beta agonist).
* History of COPD exacerbation or lower respiratory track infection that required treatment with antibiotic, oral or parenteral corticosteroid within the last 3 days prior the screening visit or during the run-in/wash-out period or history of respiratory tract infection that required treatment with antibiotic within the last 14 days prior the screening visit.
* Hospitalization due to COPD or pneumonia within the last 3 mounts prior the screening visit.
* SGOT (serum glutamic-oxaloacetic transaminase) >80 IU/L, SGPT (serum glutamic-pyruvic transaminase) >80 IU/L, bilirubin >2.0 mg/dL or creatinine >2.0 mg/dL.
* History of asthma, significant chronic respiratory diseases (i.e., significant bronchiectasis, interstitial lung diseases, etc.) other than COPD or presence of disease that may be serious and/or potentially affect results of the study.
* Use of beta-blocker, monoamine oxidase (MAO) inhibitor or tricyclic antidepressant within the last 30 days prior the screening visit
* Recent (within ≤3 months prior the screening visit) history of heart attack, heart failure, acute ischemic heart disease or presence of serious cardiac arrhythmia requiring drug treatment.
* Regularly use of daytime CPAP (continuous positive airway pressure) oxygen therapy for longer than 1 hour per day.
* Initiation of pulmonary rehabilitation within the 3 months prior the screening visit.
* History of lung volume reduction surgery
* Drug or alcohol abuse
* Presence of active tuberculosis
* History of atopy or allergic rhinitis
* Presence of active cancer
* Attenuated live virus vaccination within the last 2 weeks prior the screening visit or during the run-in/wash-out period
* Pregnancy or lactation
* Presence of known symptomatic prostatic hypertrophy requiring treatment
* Presence of known narrow-angle glaucoma requiring treatment
* Currently participating in another clinical trial or treatment with another investigational study drug within the last month or 6-half-lives, whichever is longer.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2023-08-25 (Actual); Primary Completion 2024-02-06 (Estimated); Study Completion 2024-03-06 (Estimated)

PRIMARY OUTCOMES:
FEV1 area under the curve from 0-8 h (FEV1 AUC0-8 h) | 8 hours
  Change From Baseline in Forced Expiratory Volume in one second (FEV1) Area Under the Curve (AUC) 0-8h.

SECONDARY OUTCOMES:
FEV1 area under the curve from 0-4 h (FEV1 AUC0-4 h) | 4 hours
  Change From Baseline in FEV1 AUC (0-4h).
FEV1 AUC4-6 h | 4 to 6 hours
  Change From Baseline in FEV1 AUC (4-6h).
FEV1 AUC6-8 h | 6 to 8 hours
  Change From Baseline in FEV1 AUC (6-8h).
FVC AUC0-4 h | 4 hours
  Change From Baseline in Forced Vital Capacity (FVC) AUC (0-4h).
FVC AUC4-6 h | 4 to 6 hours
  Change From Baseline in FVC AUC (4-6h).
FVC AUC6-8 sa | 6 to 8 hours
  Change From Baseline in FVC AUC (6-8h).
FVC AUC0-8 sa | 8 hours
  Change From Baseline in FVC AUC (0-8h).
Change From Baseline in FEV1 and FVC within the first 15 minutes after dosing | Baseline, 15 minutes post-dose at treatment day.
  Spirometric measurements will be performed pre-treatment and 5 min, 15 min, 30 min, 45 min and 1 h, 2 h, 3 h, 4 h, 5 h, 6h, 7h, 8h after drug administration. The measurements at the time points related to the outcome will be evaluated.
Mean Maximum Change From Baseline in FEV1 and FVC within the first 2 hours after dosing | Baseline, 2 hours post-dose at treatment day
  Spirometric measurements will be performed pre-treatment and 5 min, 15 min, 30 min, 45 min and 1 h, 2 h, 3 h, 4 h, 5 h, 6h, 7h, 8h after drug administration. The measurements at the time points related to the outcome will be evaluated.
Mean Maximum Change From Baseline in FEV1 and FVC over a period of 8 hours | Baseline, 0 to 8 hours post-dose at treatment day
  Spirometric measurements will be performed pre-treatment and 5 min, 15 min, 30 min, 45 min and 1 h, 2 h, 3 h, 4 h, 5 h, 6h, 7h, 8h after drug administration.
The Time to Onset of Bronchodilator Response | Baseline, 0 to 8 hours post-dose at treatment day
  Bronchodilator response is defined as 100 mL improvement in FEV1.
Evaluation of Safety | Baseline, 0 to 24 hours post-dose
  Number of participants with Adverse Events, with abnormal physical examinations, abnormal laboratory test results and abnormal ECGs

CONTACTS AND LOCATIONS:
Locations (1):
- Yedikule Chest Diseases And Thoracic Surgery Training And Reseaerch Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No